CLINICAL TRIAL: NCT00573807
Title: Phase 1 Study to Evaluate the Efficacy of Using Energy Specific Far Infrared Radiation Treatment for Sciatica.
Brief Title: Energy Specific Far Infrared Radiation Treatment for Sciatica
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder & President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-SCIA-CTP1
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2009-01

CONDITIONS: Sciatica
Keywords: Neuralgia, Sciatic; Sciatic Neuralgia; Sciatica, Bilateral; Lower back pain
MeSH Terms: conditions — Sciatica; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Radiation: Far Infrared Radiation (5μm to 20μm wavelength)

INTERVENTIONS:
Radiation: Far Infrared Radiation (5μm to 20μm wavelength) — Far Infrared Radiation (5μm to 20μm wavelength)for 30 to 40 minutes per treatment session.

SUMMARY:
A preliminary study to determine the use of far infrared radiation for the treatment of back pain

DETAILED DESCRIPTION:
Sciatica is created by joint misalignment, muscle spasm and inflammation. Generally, sciatica is a combination of lower back pain, pain radiating into the buttock and possibly down the leg.

Far infrared radiation of the sciatic nerve, coupled with the stretching of the spinal cord, is a promising non-invasive method for treating sciatica.

ELIGIBILITY:
Inclusion Criteria:

* Persons with lower back pain

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-03 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
The primary end point is to determine the therapeutic effects of far infrared radiation on the Sciatic nerve. | 2 years and 6 months

SECONDARY OUTCOMES:
Far infrared treatment for other pain syndromes | 2 years and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Study Director — GAAD Medical Research Institute Inc.; Kwasi Donyina, Ph.D., Study Chair — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada